CLINICAL TRIAL: NCT02406430
Title: Preoperative Prognostic Factors and Predictive Score in Patients Operated on for Combined Cataract and Idiopathic Epiretinal Membrane.
Brief Title: Prognostic Factors in Epiretinal Membrane Surgery
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: CREUZOT 2013
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Epiretinal Membranes
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

INTERVENTIONS:
Procedure: a combined cataract and ERM surgery — All patients underwent a combined cataract and ERM surgery owing to visual impairment or disabling metamorphopsia. A complete ophthalmological examination was performed before and at 1,6, and 12 months after the surgery, including best corrected visual acuity with Snellen charts converted into the logarithm of the minimum angle of resolution, slit-lamp biomicroscopy, indirect fundus, and macular optical coherence tomography

SUMMARY:
Retrospective interventional case series study reporting preoperative clinical and anatomical factors associated with visual recovery 1 year after combined cataract and idiopathic epiretinal membrane surgery. Age, duration of symptoms, and preoperative best corrected visual acuity appeared to be reliable prognostic factors. Combining these factors with analysis of the photoreceptors' inner and outer segments junction in spectral-domain optical coherence tomography provides a predictive score to estimate individual chances of good visual recovery

ELIGIBILITY:
Inclusion Criteria:

* symptomatic idiopathic epiretinal membrane operated on between April 2009 and September 2012 at the university hospital of Dijon, France.
* All patients signed informed consent for the surgical procedure.

Exclusion Criteria:

* Patients were excluded if they presented any cause of secondary epiretinal membrane (including diabetic retinopathy, vein occlusion, ocular inflammation, retinal detachment, or previously vitrectomized eye), high myopia (axial length ≥ 26 mm or spherical equivalent ≥ 6 diopters), severe media opacities with weak SD-OCT signal strengths, or any macular or optic nerve disease. Patients with a follow-up of less than 12 months were excluded and only one eye was included in those with bilateral epiretinal membranes.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated on for combined cataract and idiopathic epiretinal membrane
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2009-04; Primary Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity | 1 year after the surgery
  Best corrected visual acuity 1 year after the surgery, and preoperative factors associated with this visual outcome (age, duration of symptoms, initial best corrected visual acuity, and optical coherence tomography findings)

SECONDARY OUTCOMES:
To set up a predictive score for a >= 20/20 best corrected visual acuity | 1 year after the surgery
  To set up a predictive score for a >= 20/20 best corrected visual acuity, 1year after a combined cataract and epiretinal membrane surgery